CLINICAL TRIAL: NCT07193615
Title: Clinical Exploratory Study of YOLT-202 in the Treatment of Alpha-1 Antitrypsin Deficiency (AATD)
Brief Title: Study of YOLT-202 in the Treatment of Alpha-1 Antitrypsin Deficiency (AATD)
Acronym: AATD
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AATD-YOLT-202-001
Record Dates: First submitted 2025-07-07; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Alpha-1 Antitrypsin Deficiency (AATD)
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Dose groups: 35mg, 45mg, 55mg, TBD (During the dose-escalation process, the investigator and the sponsor may decide, based on actual circumstances, whether to add new dose groups or repeat completed dose groups for the exploratory study).
  Interventions: Drug: YOLT-202

INTERVENTIONS:
Drug: YOLT-202 — The IP is administered intravenously at the predetermined dose; Administration frequency: Once
  Other Names: AATD-YOLT-202-001

SUMMARY:
This is a single-arm, open-label, single-dose, dose-escalation exploratory study to evaluate the safety and tolerability of a single dose of YOLT-202 in patients with AATD and determine the optimal biologically active dose (OBD) of YOLT-202.

DETAILED DESCRIPTION:
This is a single-arm, open-label, single-dose, dose-escalation exploratory study to evaluate the safety and tolerability of a single dose of YOLT-202 in patients with AATD, determine the OBD of YOLT-202, and preliminarily assess the impact of a single dose of YOLT-202 on changes in FEV1 and FEV1/FVC ratio from baseline after bronchodilator use.

Note: The OBD is defined as the dose achieving either a blood functional-AAT/total-AAT protein ratio of 50%-95% at Day 21 post-dose, or a blood total-AAT protein concentration ≥ 11 μM at Day 21 post-dose. OBD ≤ maximum tolerated dose (MTD).

In this study, the maximum screening period of the main study is 60 days, the treatment day is D0, and the safety follow-up period is up to Week 52 after administration. In the main study, when OBD is achieved, additional subjects will be added to the dose group (the sponsor and the investigator will jointly negotiate the specific number of subjects) for further verification. After completing safety follow-up, subjects may voluntarily receive a second dose of the investigational drug at the OBD level based on comprehensive assessments of efficacy, safety, and PK/PD data.

After the end of the main study, the subjects will undergo long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (inclusive) aged ≥ 18 and ≤ 70 years old at the time of signing informed consent.
* Diagnosed with AATD and genetically confirmed as homozygous PiZZ mutation.
* Blood total AAT level < 11 μM or equivalent protein in mg/dL.
* Patients receiving augmentation therapy must be willing to discontinue it at least 6 weeks prior to signing the informed consent form (ICF) and throughout the study period, unless clinically indicated.

Exclusion criteria

* Body mass index (BMI) > 35 kg/m2.
* Patients who have undergone lung or liver transplantation, are on the waiting list for lung or liver transplantation, or have had lung volume reduction surgery (LVRS).
* Clinical evidence of severe bronchiectasis, as judged by the investigator (e.g., excessive sputum production or recurrent infections requiring antibiotics [> 4 times per year]).
* FEV1 ≤ 30% of predicted value after bronchodilator use at screening
* Liver disease with any of the following:

  * Measured liver stiffness (FibroScan) ≥ 10 kilopascals (kPa).
  * Known history of hepatic cirrhosis or associated complications (e.g., varices, ascites, hepatic encephalopathy).
  * ≥ F2 hepatic fibrosis in patients with prior liver biopsy.
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times the upper limit of normal (ULN).
  * Total bilirubin > ULN; or > 2 times the ULN if Gilbert's syndrome is documented.
  * International normalized ratio (INR) ≥ 1.2 at screening. If deemed appropriate by the investigator and/or the prescribing physician, anticoagulants may be discontinued for a washout period or reversed with vitamin K. If necessary, a repeat INR < 1.2 is acceptable.
  * Hepatitis B surface antigen (HBsAg) positive.
  * Hepatitis C virus (HCV) antibody positive. If HCV antibody is positive, HCV RNA PCR must be negative.
* Allergy to the drugs contained in lipid nanoparticles (LNP) or LNP-mRNA vaccines, or previous history of adverse reactions to LNP-based drugs;
* Smoking more than 5 cigarettes per day or consuming the equivalent amount of nicotine or nicotine replacement products within the past 6 months before screening.
* History of alcohol abuse within the past 6 months before screening (drinking more than 14 units of alcohol per week [1 unit ≈ 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine]); or positive alcohol breath test at the time of screening or admission.
* Patients with poorly controlled hypertension by conventional treatments (systolic blood pressure [SBP] ≥ 180 mmHg and/or diastolic blood pressure [DBP] ≥ 110 mmHg).
* Patients with poorly controlled diabetes (hemoglobin A1c ≥ 9%).
* Presence of New York Heart Association (NYHA) class III-IV heart failure, left ventricular ejection fraction < 50%, or prolonged QTc interval (female > 470 ms, male > 450 ms) at the time of screening.
* Myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, coronary artery bypass grafting, severe deep vein thrombosis or pulmonary embolism within 3 months before screening; poorly controlled severe arrhythmias within the past 3 months before screening, such as poorly controlled recurrent and highly symptomatic ventricular tachycardia, rapid ventricular response atrial fibrillation, or supraventricular tachycardia; or planned cardiac surgery or cardiac revascularization during the main study period.
* Cerebrovascular accidents within 6 months before screening;
* Known or suspected systemic viral, parasitic, or fungal infections, or active infections requiring expected antibiotic therapy within 14 days after screening.
* Human immunodeficiency virus (HIV) antibody positive at screening.
* Anticoagulant therapy within 14 days before enrollment (such as warfarin, dabigatran, apixaban).
* Patients with bleeding tendency or history of coagulation disorders (such as liver cirrhosis, malignant hematological diseases, antiphospholipid antibody syndrome);
* Expected survival time less than 2 years.
* History of malignant tumors within the past 5 years (excluding cured skin basal cell carcinoma, skin squamous cell carcinoma, cervical carcinoma in situ, low-grade prostate carcinoma in situ, and cured thyroid basal cell carcinoma).
* History of drug abuse within the past 3 years.
* Pregnant or lactating women.
* Patients with other diseases in the blood system, digestive system, central nervous system, or endocrine system that the investigator believes will interfere with evaluation or limit participation in the trial.
* Inability or unwillingness to cooperate or comply with pretreatment medication requirements or study procedures.
* Any other condition deemed unsuitable for the clinical trial participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety of YOLT-202 in subjects after administration | Baseline to 52 weeks post-dose
  Numbers and percentages of patients with adverse events (AE)

SECONDARY OUTCOMES:
Pharmacokinetics parameter of YOLT-202 | 30 minutes pre-dose, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 168 hours, 336 hours and 504 hours post-dose
  Post-dose plasma concentration (Cmax)
Pharmacokinetic (PK) parameter of YOLT-202 | 30 minutes pre-dose, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 168 hours, 336 hours and 504 hours post-dose
  Evaluate the time of maximum concentration (tmax)
Pharmacokinetic (PK) parameter of YOLT-202 | 30 minutes pre-dose, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours, 168 hours, 336 hours and 504 hours post-dose
  To evaluate the area under curve (AUC)
Pharmacokinetic (PK) parameters of YOLT-202 | 30 minutes pre-dose, 2 hours, 6 hours, 24 hours, 48 hours, 72 hours,168 hours,336 hours and 504 hours post-dose
  To evaluate elimination half-life (t1/2)
Changes in blood AAT protein level | Weeks 1, 2, 3 and 52 post-dose
  Total -AAT level over time

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No